CLINICAL TRIAL: NCT04458064
Title: I-gel Versus Air-Q LMA for Pediatric Patients Undergoing Short-duration Surgical Procedures
Brief Title: I-gel Versus Air-Q LMA for Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ayman Anis Metry, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASUH1421/18
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Easy Insertion, Complications Ans Suitability of i Gel and Air Q LMA

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i gel (Active Comparator): I gel LMA was inserted for all patients
  Interventions: Other: LMA i gel
- Air Q LMA (Active Comparator): Air Q LMA was inserted for all patients
  Interventions: Other: LMA i gel

INTERVENTIONS:
Other: LMA i gel — insertion of LMA for maintaining airway during anesthesia
  Other Names: LMA Air Q

SUMMARY:
This study targets to compare insertion facility, effect on hemodynamic parameters and effective ventilation using i-gel versus Air-Q LMA for pediatric patients undergoing short-duration surgical procedures.

DETAILED DESCRIPTION:
The patient were divided into 2 groups. I gel group and Air Q group according to LMA type used to maintain airway ventilation.

The patients were compared according to insertion facility, effect on hemodynamic parameters and effective ventilation.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I-II
* operative time of ≤60 minutes

Exclusion Criteria:

* age >10 years
* ASA grade ≥II
* current or recently resolved upper respiratory tract infection
* presence of oropharynx or laryngeal pathologies or congenital anomalies
* pathologies inducing reflux or increasing the possibility of aspiration
* allergy to anaesthetic or drugs to be used, renal, cardiac or hepatic diseases, or bronchial asthma

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Supraglottic device success rate | 60 minutes
  Fitness of LMA for ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt